CLINICAL TRIAL: NCT04957277
Title: Stepping to Understand Lower Limb Impairments in Bilateral Cerebral Palsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Theresa Moulton, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00214804
Record Dates: First submitted 2021-06-28; First posted 2021-07-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy; Bilateral Cerebral Palsy; Diplegic Cerebral Palsy
Keywords: Cerebral Palsy; Bilateral Cerebral Palsy; Gait; Stepping; Stairs; Biomechanics; Neuroscience
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: All participants are exposed to all conditions in a randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- load modulation (Experimental): Participants will experience different body weight loading conditions - with body weight added by a weighted vest or removed using the ZeroG overhead harness.
  Interventions: Other: load modulation

INTERVENTIONS:
Other: load modulation — Adding body weight (BW) up to 20% BW and subtracting body weight down to -20% BW

SUMMARY:
The purpose of this study is to investigate lower limb impairments in children with bilateral cerebral palsy during stepping tasks.

DETAILED DESCRIPTION:
Individuals with bilateral cerebral palsy (BCP) sustain a neonatal brain injury that leads to altered neuromuscular control to the lower limbs. One commonly observed motor impairment from this altered control is loss of selective voluntary motor control (SVMC), defined as the ability to independently move the joints intentionally. Loss of SVMC typically manifests as knee and ankle joint impairment and abnormal coupling between the hip adductors and lower limb extensors. This can make stepping up or down a curb or stair challenging, but quantitative investigation in these closed-chain activities has been limited. This is especially important as performance in stair-climbing is associated with limitations to overall mobility and community participation in cerebral palsy.

The overall aim of this proposal is to investigate the altered neuromuscular control that challenges stair walking in individuals with BCP. Participants who consent to the study will be instructed to perform multiple step-ups and step-downs on a single raised platform. The parameters of the stepping task may change by adding weight to the body or subtracting weight from the body. Using standard gait analysis techniques, biomechanical metrics such as joint kinematics and kinetics will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* aged 5 years to 19 years
* typically developing with no diagnosed medical conditions that affect movement, OR with a diagnosis of bilateral cerebral palsy (including diplegia, tetraplegia, and quadriplegia) where the lower limbs are more affected than the upper limbs
* ability to independently step up, with or without assistive devices.

Exclusion Criteria:

* lower limb surgery in the past year
* botulinum toxin injections to the lower limb muscles in the past 6 months
* cognitive dysfunction that would make following directions difficult
* comorbidities that would make participation unsafe.

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Joint biomechanics (support moment) | At baseline and each loading level; During entirety of the stepping trial, from initial lift-off to final contact onto the single platform.
  Sum of the joint kinetics from the hip, knee and ankle, termed the "support moment" and measured in Nm.
Joint biomechanics (hip) | At baseline and each loading level; During entirety of the stepping trial, from initial lift-off to final contact onto the single platform.
  hip torque (measured in Nm) will be identified for the hip, knee, and ankle during the duration of the task.
Joint biomechanics (knee) | At baseline and each loading level; During entirety of the stepping trial, from initial lift-off to final contact onto the single platform.
  Knee angle (between the thigh and shank measured in degrees) will be identified during the duration of the task.
Joint biomechanics (ankle) | At baseline and each loading level; During entirety of the stepping trial, from initial lift-off to final contact onto the single platform.
  Ankle angle (between the shank and foot measured in degrees) will be identified during the duration of the task.

SECONDARY OUTCOMES:
Muscle activations (hip) | At baseline and each loading level; During entirety of the stepping trial, from initial lift-off to final contact onto the single platform.
  EMG data will be identified for underlying muscles of the hip during the stance phases of the task.
Muscle activations (knee) | At baseline and each loading level; During entirety of the stepping trial, from initial lift-off to final contact onto the single platform.
  EMG data will be identified for underlying muscles of the knee during the stance phases of the task.
Muscle activations (ankle) | At baseline and each loading level; During entirety of the stepping trial, from initial lift-off to final contact onto the single platform.
  EMG data will be identified for underlying muscles of the ankle during the stance phases of the task.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw data files underlying publications will be shared
Time Frame: Upon publication
URL: https://arch.library.northwestern.edu/?locale=en

REFERENCES:
- [Background] Rose J. Selective motor control in spastic cerebral palsy. Dev Med Child Neurol. 2009 Aug;51(8):578-9. doi: 10.1111/j.1469-8749.2009.03401.x. No abstract available. PMID 19627331
- [Background] Fowler EG, Staudt LA, Greenberg MB. Lower-extremity selective voluntary motor control in patients with spastic cerebral palsy: increased distal motor impairment. Dev Med Child Neurol. 2010 Mar;52(3):264-9. doi: 10.1111/j.1469-8749.2009.03586.x. PMID 20089048
- [Background] Novak AC, Brouwer B. Sagittal and frontal lower limb joint moments during stair ascent and descent in young and older adults. Gait Posture. 2011 Jan;33(1):54-60. doi: 10.1016/j.gaitpost.2010.09.024. Epub 2010 Oct 30. PMID 21036615
- [Background] Lepage C, Noreau L, Bernard PM. Association between characteristics of locomotion and accomplishment of life habits in children with cerebral palsy. Phys Ther. 1998 May;78(5):458-69. doi: 10.1093/ptj/78.5.458. PMID 9597060